CLINICAL TRIAL: NCT06771362
Title: Evaluation of ART Restorations Using Two Different Bulk-Fill Restorative Materials in Primary Molars With 12-month Follow-up According to Modified USPHS and Revised FDI Criteria
Brief Title: Evaluation of ART Restorations Using Two Different Bulk-Fill Restorative Materials in Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Idil Ay Simsek, Research Assistant, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMU-FD-PD-IASIMSEK-001
Record Dates: First submitted 2025-01-06; First posted 2025-01-13 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Dentin Caries
Keywords: tooth demineralization; dental caries; Stomatognathic Diseases; Atraumatic Restorative Treatment
MeSH Terms: conditions — Tooth Demineralization; Dental Caries; Stomatognathic Diseases | interventions — glass ionomer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STELA BULK-FILL RESTORATION (Experimental): Stella Bulk-Fill composite restoration after ART
  Interventions: Procedure: ART with Bulk-Fill composite
- GLASS IONOMER (Control) (Other): RIVA Self-Cure HV glass ionomer restoration after ART
  Interventions: Procedure: ART with Glass Ionomer

INTERVENTIONS:
Procedure: ART with Bulk-Fill composite — Restoration using Bulk-fill flowable self-cured composite
  Arms: STELA BULK-FILL RESTORATION
Procedure: ART with Glass Ionomer — Restoration Using High-Viscosity Glass Ionomer Cement
  Arms: GLASS IONOMER (Control)

SUMMARY:
The aim of this clinical study is to evaluate the success of two different bulk-fill restorative materials applied to teeth restored with atraumatic treatment at 3, 6, and 12-month follow-ups. The research seeks to address the following questions:

Which bulk-fill restorative material is more effective in terms of clinical success? How does the clinical success of bulk-fill restorations change over time (3, 6, and 12 months)? How do the two materials compare in terms of functional, aesthetic, and biological outcomes? To what extent does the cavity size of teeth with interproximal caries, restored using atraumatic treatment, influence treatment success? In this study, asymptomatic teeth with aproximal caries in children aged 4-9 will be repaired using atraumatic treatment and assessed based on the Modified USPHS (United States Public Health Service) and Revised FDI (World Dental Federation) criteria.

DETAILED DESCRIPTION:
Atraumatic Restorative Treatment (ART) is a minimally invasive approach developed for treating dental caries. This method involves removing carious tissue to the minimum extent possible using hand instruments and restoring the cavity with a biocompatible material, such as high-viscosity glass ionomer cement (GIC). The fundamental principle of ART is to preserve the tooth's natural structure while providing a more comfortable and accessible treatment for patients. It offers a less stressful experience, particularly for children or patients with dental anxiety.

Patients between the ages of 4-9 who meet ICDAS II (International Caries Detection and Assessment System) 4-5-6 criteria and need restoration of asymptomatic primary molars with unilateral or multifaceted carious cavities will be included. Volunteers will be randomly divided into two groups, and the treatments of primary molars will be completed using two different high-viscosity glass ionamer cement (HV-GIC). The teeth in all groups will be cleaned of decay using an excavator down to the affected dentin. After the cavity is prepared, the tooth is isolated using cotton pellets.

Group 1: (RIVA Self Cure/HV, SDI, Australia) Apply a dentin conditioner (Riva Conditioner, SDI, Australia) to the prepared dentin surface for 10 seconds, then rinse thoroughly with water and gently blot dry. Ensure the tooth surface remains moist. The tooth will be restored with RIVA Self Cure (SDI, Australia) capsule form by the manufacturer's instructions, and the restoration will be covered with a sealing agent (RIVA Coat, SDI, Australia) Group 2: (STELA , SDI, Australia) STELA Primer (SDI, Australia) to the prepared cavity surface using a disposable brush applicator and leave it for 5 seconds. After drying the teeth, place the syringe into the mixer and follow the manufacturer's instructions for mixing. Apply the mixed STELA restorative material directly into the prepared cavity. The restoration is completed following the manufacturer's recommendations.

Before the procedure, demographic and dental data of the child volunteer, such as age, gender, brushing frequency, and number of teeth treated, will be recorded.

The US Public Health Service criteria (retention, anatomical form, surface roughness, secondary caries, marginal discoloration, and marginal integrity) and Modified FDI criteria will be used for clinical evaluation of restorations. The restorations will be evaluated clinically and radiologically at baseline 3., 6. and 12. months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients and parents of the patients who accept to participate and sign the informed consent.
2. Children between the ages of 4-9
3. Healthy children without a history of serious systemic conditions necessitating chronic use of medications.
4. Children whose dental examination reveals at least one untreated asymptomatic cavitated carious lesion (ICDAS II index: code 4,5,6) affecting primary molars.
5. Absence of former history of spontaneous pain from the offending tooth/teeth.
6. Patients with an appropriate level of cooperation to complete treatment under clinical conditions.
7. Teeth are in a restorable condition. Natural exfoliation of primary teeth to be treated should not be expected within two years.

Exclusion Criteria:

1. Patients and parents of the patients who does not accept to participate and sign the informed consent
2. Patients with special health care needs or any medical conditions.
3. Primary molar teeth with excessive crown damage that cannot be restored.
4. Primary molar teeth in which bone loss exceeds 1/3 of the roots.
5. Primary molar teeth that have previously undergone root canal treatment or pulpotomy treatment.
6. Presence of internal/external and root resorption in primary teeth to be treated.
7. Root fracture, ankylosis or mobility in the primary teeth to be treated.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Change form 3 months to 12 months regarding | 3-month,6-month,12 month
  alpha: The general contour of the restorations follows the contour bravo: the general contour of the restoration does not follow the contour of the tooth charlie: The restoration has an overhang does
Change from 3 months to 12 months regarding "Marginal adaptation" | 3-month,6-month,12 month
  alpha: Explorer does not catch or has one-way catch when drawn across the restoration/tooth interface bravo: explorer falls into crevice drawn across the restoration/tooth interface charlie: Dentin or base is exposed along the margin
Change from 3 months to 12 months regarding "Surface roughness" | 3-month,6-month,12 month
  alpha: the surface of the restoration does not have any surface defects bravo: the surface of the restoration has minimal surface defects charlie: the surface of the restoration has severe surface defects
Change from 3 months to 12 months regarding "Marginal staining" | 3-month,6-month,12 month
  alpha: there is no discoloration between the restorations and tooth bravo: there is discoloration on less than half of the circumferential margin charlie: there is discoloration on more than half of the circumferential margin
Change from 3 months to 12 months regarding "Retention" | 3-month,6-month,12 month
  alpha: intact bravo: chipped/loss of material charlie: complete loss of crown
Change from 3 months to 12 months regarding "Incisal wear" | 3-month,6-month,12 month
  alpha: intact bravo: wear of occlusal surface without tooth surface exposure charlie: wear of occlusal surface with tooth surface exposure
Functional properties according to revised FDI (World Dental Federation) criteria. | 3-month,6-month,12 month
  Functional properties:
  F2: Marginal adaptation measured by visual examination, short air drying, 250 μm probe.
  F3:Proximal contact point measured by visual examination and 25/50/100 μm blades.
  F4: Form and contour measured by visual examination. F5: Occlusion and occlusal wear measured by visual examination and articulation paper.
  Method of aggregation is frequency and percentage. Measuring unit is scoring system (Ordinal, scores 1-5). (1) Clinically excellent. (sufficient). (5) Clinically poor (entirely insufficient).
Biological properties according to revised FDI criteria | 3-month,6-month,12 month
  Biological properties:
  B1: Caries at restoration margin (CAR) measured by visual examination, short air drying, and 250 μm probe.
  B2: Dental hard tissue defects at restoration margin measured by visual examination.
  B3: Postoperative hypersensitivity reported by patient and pulp status tested with cold stimulus.
  Method of aggregation is frequency and percentage. Measuring unit is scoring system (Ordinal, scores 1-5). (1) Clinically excellent. (sufficient). (5) Clinically poor (entirely insufficient).
Aesthetic properties according to revised FDI criteria | 3-month,6-month,12 month
  Aesthetic properties:
  A1: Surface luster and surface texture measured by visual examination and short air drying.
  A2: Marginal staining measured by visual examination and short air drying. A3: color match measured by visual examination. Method of aggregation is frequency and percentage. Measuring unit is scoring system (Ordinal, scores 1-5). (1) Clinically excellent. (sufficient). (5) Clinically poor (entirely insufficient).

CONTACTS AND LOCATIONS:
Locations (1):
- Canakkale Onsekiz Mart University, Çanakkale, Kepez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In this study, the investigators are committed to sharing our findings while ensuring the privacy and confidentiality of our participants. Therefore, the investigators will only be disseminating aggregated statistical results derived from the data, rather than individual participant data.